CLINICAL TRIAL: NCT01030068
Title: Yoga for Women Attempting Smoking Cessation: An Initial Investigation
Brief Title: Yoga for Smoking Cessation Feasibility Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: The Miriam Hospital (Other)
Collaborators: Rhode Island Hospital (Other); Brown University (Other)
Responsible Party: Principal Investigator, Beth Bock, Ph.D., Professor of Psychiatry & Human Behavior, The Miriam Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: R21AT003669 (NIH)
Record Dates: First submitted 2009-12-09; First posted 2009-12-11 (Estimated); Last update posted 2011-10-07 (Estimated); Status verified 2011-10

CONDITIONS: Smoking Cessation
Keywords: Smoking Cessation; Yoga; Wellness; Feasibility; Smoking Cessation Therapy
MeSH Terms: conditions — Smoking Cessation | interventions — Yoga; Health

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Yoga (Experimental): Yoga plus smoking cessation
  Interventions: Behavioral: Yoga; Other: Smoking cessation therapy
- Wellness (Active Comparator): Health & Wellness classes plus smoking cessation therapy
  Interventions: Behavioral: Wellness; Other: Smoking cessation therapy

INTERVENTIONS:
Behavioral: Yoga — Yoga twice weekly
  Arms: Yoga
Behavioral: Wellness — Health and wellness classes twice weekly
  Arms: Wellness
Other: Smoking cessation therapy — Smoking cessation therapy

SUMMARY:
The purpose of this study is to test whether it is feasible to provide a smoking cessation program together with a yoga program to help women quit smoking. We anticipate that women will be enthusiastic about the program and that we will be able to recruit and treat women for smoking cessation within the designated time frame.

DETAILED DESCRIPTION:
Cigarette smoking is the leading preventable cause of morbidity and mortality among adults in the United States. Smoking, and quitting smoking may be especially problematic for women. Our prior research has demonstrated that traditional aerobic exercise (e.g., brisk walking, bicycling) improves cessation outcomes among women. Exercise appears to reduce the effects of nicotine withdrawal and improves cessation outcomes by improving mood and reducing weight gain. yoga that shares many of the same properties of the traditional aerobic exercise that has been shown to be an efficacious adjunct to smoking cessation treatment. Moreover, some features of yoga, including a focus on breathing, meditation, stress reduction and enhanced mood are likely to have special relevance to smokers who are trying to quit. Thus, yoga may prove to be a more efficacious complimentary treatment for smoking cessation than traditional aerobic exercise.

The goal of this proposal is to conduct an initial investigation of the efficacy of providing Yoga as an adjunct to cognitive behavioral treatment (CBT) for smoking cessation. Adult women smokers (n=72) will be recruited through newspaper advertisements and will be randomly assigned to either: (1) CBT plus Yoga , or (2) CBT plus contact control. All study participants will be given a sub-maximal exercise stress test to ensure that they are safe to exercise. Yoga sessions will be conducted twice weekly for 12 weeks, and will be lead by certified instructors in yoga. Smoking cessation sessions will be conducted once per week for 12 weeks and will be lead by Masters or PhD level specialists in smoking cessation. Differences in post-treatment (12 week) cessation rates (7-day point prevalence abstinence) will provide data for estimates of effect size between conditions. This effect size estimate is necessary in order to calculate power estimates for a major clinical trial.

ELIGIBILITY:
Inclusion Criteria:

* healthy female smokers
* ages 18-65
* smoke 10+ cigarettes a day
* sedentary (not exercising more than 2 times per week)

Exclusion Criteria:

* major depression
* hypertension
* more than 1 year previous yoga experience
* current experience with yoga or smoking cessation treatment

Ages: 18 Years to 65 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2007-07; Primary Completion 2011-07 (Actual); Study Completion 2011-07 (Actual)

PRIMARY OUTCOMES:
Recruitment and qualitative feasibility | 10 week

SECONDARY OUTCOMES:
Smoking cessation | 6 month

CONTACTS AND LOCATIONS:
Overall Officials: Beth C Bock, PhD, Principal Investigator — The Miriam Hospital
Locations (1):
- The Miriam Hospital, Providence, Rhode Island, United States